CLINICAL TRIAL: NCT02269085
Title: A Phase I/II Trial of Ibrutinib (BTK Inhibitor) in Combination With Carfilzomib in Relapse/Refractory Mantle Cell Lymphoma
Brief Title: Trial of PCI-32765 (BTK Inhibitor) in Combination With Carfilzomib in Relapse/Refractory Mantle Cell Lymphoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: slow accrual
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Pharmacyclics LLC. (Industry); Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013-0677; NCI-2014-02495 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2014-10-16; First posted 2014-10-20 (Estimated); Last update posted 2019-02-28 (Actual); Status verified 2019-02

CONDITIONS: Lymphoma
Keywords: Lymphoma; Mantle cell lymphoma; MCL; Relapsed or refractory; Ibrutinib; PCI-32765; Imbruvica; Carfilzomib
MeSH Terms: conditions — Lymphoma; Lymphoma, Mantle-Cell; Recurrence | interventions — ibrutinib; carfilzomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ibrutinib + Carfilzomib (Experimental): Phase I: Ibrutinib administered by mouth daily at 420 or 560 mg on Days 1 - 28 of a 28-day cycle. Carfilzomib administered by vein 20/27 mg/m^2, 20/36 mg/m^2, 20/45 mg/m^2 or 20/56 mg/m^2 on days 1, 2, 8, 9, 15 and 16 of a 28-day cycle for Cycles 1- 12 and on Days 1, 2, 15 and 16 for Cycle 13 and higher.
  Phase II: Once the MTD has been established 5 additional patients treated at the MTD to a maximum of 35 patients with MCL.
  Study staff calls participant after end-of-dosing visit every 6 months for 5 years.
  Interventions: Drug: Ibrutinib; Drug: Carfilzomib; Behavioral: Phone Calls

INTERVENTIONS:
Drug: Ibrutinib — Phase I Starting Dose: 420 mg by mouth daily on Days 1 - 28 of a 28-day cycle.
  Phase II Starting Dose: MTD from Phase I.
  Other Names: PCI-32765; Imbruvica
Drug: Carfilzomib — Phase I Starting Dose: 20 mg/m2 by vein on Days 1, 2, 8 ,9, 15 and 16 in Cycles 1 - 12, and Days 1,2 and 15,16 of Cycle 13 and beyond.
  Phase II Starting Dose: MTD from Phase I.
Behavioral: Phone Calls — Study staff calls participant after end-of-dosing visit every 6 months for 5 years. These calls should take about 2-3 minutes.

SUMMARY:
The goal of this clinical research study is to find the highest tolerable dose of carfilzomib and ibrutinib that can be given to patients with relapsed or refractory MCL.

Researchers also want to learn if carfilzomib and ibrutinib can help to control the disease.

This is an investigational study. Ibrutinib is FDA approved and commercially available to treat MCL and chronic lymphocytic leukemia (CLL). Carfilzomib is FDA approved and commercially available to treat certain types of multiple myeloma. Giving carfilzomib to patients with MCL is investigational. The combination of ibrutinib and carfilzomib is investigational. The study doctor can explain how the study drugs are designed to work.

Up to 35 participants will be enrolled on this study. All will be enrolled at MD Anderson.

DETAILED DESCRIPTION:
Study Drug Administration:

If you are found to be eligible for this study, you will begin the first cycle of ibrutinib and carfilzomib. Each cycle is 28 days.

Ibrutinib Dosing:

You will take 2-4 ibrutinib capsules (depending on when you enter the study) every day with 1 cup (about 8 ounces) of water. The number of capsules will depend on when you enter the study. You must take all capsules at about the same time every day, at least 30 minutes before eating or at least 2 hours after a meal. Do not open the capsules or dissolve them.

If you miss a dose, you can take it up to 6 hours after the time you would have taken it. If it is later than 6 hours, you should skip the dose and start taking the capsules at the same time as usual the next day.

If you vomit a dose and can see all of the capsules you took, you can retake the dose. If you vomited and cannot see all of the capsules, do not retake the dose. Start taking the capsules at the same time as usual the next day.

You will need to fill out diary cards with information about when you take ibrutinib. You should bring the diary cards with you to every visit.

Carfilzomib Dosing:

On Days 1, 2, 8, 9, 15, and 16 of Cycles 1-12, you will receive carfilzomib by vein over about 30 minutes. The first 2 doses you receive may be lower than later doses. This is to lower the risk of an allergic reaction.

On Days 1, 2, 15, and 16 of Cycles 13 and beyond, you will receive carfilzomib by vein over about 30 minutes.

You should drink at least 6-8 cups (8 ounces each) of water or other fluids per day, starting 2 days before your first dose and for as long as your doctor asks you to. During Cycle 1, you will receive fluids by vein before your dose of carfilzomib. If your doctor thinks it is needed, you will also receive fluids by vein before each dose of carfilzomib in Cycle 2.

Before you receive carfilzomib, you will be given standard drugs to help decrease the risk of side effects. You may ask the study staff for information about how the drugs are given and their risks.

During Cycle 1 and on Day 1 of Cycle 2, you will be checked for side effects for 1 hour after you receive carfilzomib.

Study Visits:

On Day 1 of all cycles:

* You will have a physical and neurological exam.
* You will have an EKG to check your heart function.
* Blood (about 2 tablespoons) will be drawn for routine tests and to see how well your blood clots.
* If your doctor thinks it is needed, you will have a PET scan to check the status of the disease.
* If your doctor thinks it is needed, you will have a bone marrow biopsy and aspiration to check the status of the disease.
* If you are able to become pregnant, blood (about 1½ tablespoons) or urine will be collected for a pregnancy test.

On Days 2, 9, and 16 of Cycles 1 and 2, blood (about 2 tablespoons) will be drawn for routine tests and to see how well your blood clots.

On Day 1 of Cycles 2, 4, and every other cycle after that until Cycle 12 and then every 3 cycles after that, you will have a CT scan to check the status of the disease.

On Day 1 of Cycles 1, 4, and every 3 cycles after that:

* You will have an EKG.
* You will have an ECHO or MUGA scan.

On Days 8 and 15 of Cycles 1 - 3:

* You will have a physical exam (Cycle 1 and Day 15 of Cycles 2 and 3 only).
* Blood (about 2 tablespoons) will be drawn for routine tests (Cycles 1 and 2, and Day 15 of Cycle 3 only).

On Day 22 of Cycle 1:

* You will have a physical exam.
* Blood (about 2 tablespoons) will be drawn for routine tests and to see how well your blood clots.

On Day 28 of Cycle 1:

* You will have an EKG.
* You will have an ECHO or MUGA scan.

If the study doctor thinks the disease has completely responded to the study treatment, the following tests and procedures will be performed to confirm the status of the disease:

You will have a colonoscopy, including a biopsy of any abnormal growths. To collect this biopsy, small amounts of tissue are removed with a cutting tool.

You will have a bone marrow biopsy. If the doctor thinks it is needed, you will have a PET scan.

The tests may be repeated any time the doctor thinks it is needed.

Length of Study:

You may continue taking the study drugs for as long as the doctor thinks it is in your best interest. You will no longer be able to take the drugs if the disease gets worse, if intolerable side effects occur, or if you are unable to follow study directions.

Your participation on the study will be over once you have completed the long-term follow-up phone calls.

End-of-Dosing Visit:

Within about 30 days after you finish taking the study drugs:

* You will have a physical and neurological exam.
* You will have an EKG to check your heart function.
* Blood (about 3-5 tablespoons) will be drawn for routine tests and to see how well your blood clots.
* You will have a PET scan and chest x-ray to check the status of the disease.
* If your doctor thinks it is needed, you will have a CT scan to check the status of the disease.
* If your doctor thinks it is needed, you will have a bone marrow biopsy and/or aspiration to check the status of the disease.
* If your doctor thinks it is needed, you will have a colonoscopy and GI endoscopy to look for abnormal areas.
* If you are able to become pregnant, blood (about 1½ tablespoons) or urine will be collected for a pregnancy test.

Long Term Follow-Up:

After your end-of-dosing visit, the study staff will call you every 6 months for 5 years to ask how you are doing and to find out about any other treatments you have received. These calls should take about 2-3 minutes. In addition to the phone calls, your medical records may be reviewed during this time as well.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have a confirmed diagnosis of mantle cell lymphoma with positivity in tissue biopsy.
2. Patients must have previously treated relapsed and/or refractory MCL with at least 2 prior lines of therapy (prior carfilzomib, ibrutinib, bortezomib, anthracycline, rituximab or stem cell transplant are acceptable). There is no upper limit for prior lines of therapy.
3. Understand and voluntarily sign an institutional review board (IRB)-approved informed consent form.
4. Age >/= 18 years at the time of signing the informed consent.
5. Patients must have bi-dimensional measurable disease (Measureable disease by CT scan defined as at least 1 lesion that measures =/>1.5 cm in single dimension.) Patient with leukemia phase (peripheral blood involvement), non-measurable disease, gastrointestinal (GI) MCL, or bone marrow (BM) MCL are also eligible.
6. Gastrointestinal or bone marrow or spleen only patients are allowable and will be analyzed separately.
7. Eastern Cooperative Oncology Group (ECOG) performance status of 2 or less
8. Serum bilirubin <1.5 mg/dl and creatinine (Cr) Clearance >/= 30 mL/min, platelet count >75,000/mm^3 and absolute neutrophil count (ANC) > 1,500/mm^3, aspartate aminotransferase (AST)/serum glutamic oxaloacetic transaminase (SGOT) and alanine aminotransferase (ALT)/serum glutamic pyruvic transaminase (SGPT) < 3 x upper limit of normal or < 5 x upper limit of normal if hepatic metastases are present. (Patients who have bone marrow infiltration by MCL are eligible if their ANC is >/= 1000/mm^3 [growth factor not allowed] or their platelet level is >/= 50,000/mm^3).
9. Willing and able to participate in all study related procedures and therapy including swallowing capsules without difficulty.
10. Females of childbearing potential (FCBP)* must have a negative serum or urine pregnancy test and must be willing to use acceptable methods of birth control during the study and for 30 days after the last dose of study treatment. * A female of childbearing potential is a sexually mature woman who: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months).
11. Male patients must use an effective barrier method of contraception during the study and for 30 days following the last dose of study treatment if sexually active with a female of childbearing potential.

Exclusion Criteria:

1. Any serious medical condition including but not limited to, uncontrolled hypertension, uncontrolled diabetes mellitus, uncontrolled infection, active/symptomatic coronary artery disease, chronic obstructive pulmonary disease (COPD), renal failure, active hemorrhage, or psychiatric illness that, in the investigators opinion places the patient at unacceptable risk and would prevent the subject from signing the informed consent form.
2. Pregnant or breastfeeding females.
3. Use of any standard/experimental anti-lymphoma drug therapy, including steroids, within 3 weeks of initiation of the study or use of any experimental non-drug therapy (e.g., donor leukocyte/mononuclear cell infusions) within 56 days of initiation of the study drug treatment.
4. Prior allogeneic stem cell transplant (SCT) within 16 weeks or autologous SCT within 8 weeks of initiation of therapy. (Patients that require immunosuppressive therapy are not eligible within 60 days of therapy.)
5. Known human immunodeficiency virus (HIV) infection. Patients with active Hepatitis B infection (not including patients with prior Hepatitis B vaccination; or positive serum Hepatitis B antibody). Hepatitis C infection is allowed as long as there is no active disease and is cleared by GI consultation.
6. All patients with central nervous system lymphoma.
7. Significant neuropathy (Grades 3-4, or Grade 2 with pain) within 14 days prior to enrollment.
8. Known history of allergy to Captisol® (a cyclodextrin derivative used to solubilize carfilzomib).
9. Contraindication to any of the required concomitant drugs or supportive treatments or intolerance to hydration due to preexisting pulmonary or cardiac impairment including pleural effusion requiring thoracentesis or ascites requiring paracentesis.
10. Malabsorption syndrome, disease significantly affecting gastrointestinal function, or resection of the stomach or small bowel or ulcerative colitis, symptomatic inflammatory bowel disease, or partial or complete bowel obstruction, or any other gastrointestinal condition that could interfere with the absorption and metabolism of ibrutinib.
11. Major surgery within 4 weeks of initiation of therapy.
12. Requires anticoagulation with warfarin or equivalent vitamin K antagonist.
13. Requires treatment with strong CYP3A inhibitors.
14. The patient has a prior or concurrent malignancy that in the opinion of the investigator, presents a greater risk to the patient's health and survival, than of the MCL, within the subsequent 6 months at the time of consent. Investigator discretion is allowed.
15. Patients with New York Heart Association (NYHA) Class III and IV heart failure, myocardial infarction in the preceding 6 months, and significant conduction abnormalities, including but not limited to atrial fibrillation, 2nd degree AV block type II, 3rd degree block, Torsade de pointe, QT prolongation (QTc > 450 msec, sick sinus syndrome, ventricular tachycardia, symptomatic bradycardia (heart rate < 50 bpm), hypotension, light headedness and syncope. Patients with atrial fibrillation will be excluded even if they are rate-controlled. If there are any active cardiac issues, cardiology consultation will be obtained for clearance.
16. Known history of Pulmonary Hypertension
17. If the left ventricular ejection fraction (LVEF) < 40, patients will be excluded.
18. Known history of Cardiomyopathy
19. Acute infection requiring treatment (systemic antibiotics, antivirals, or antifungals) within 14 days prior to initiation of study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2015-04-20 (Actual); Primary Completion 2018-05-29 (Actual); Study Completion 2018-05-29 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of Carfilzomib When Given With Ibrutinib | 28 days
  MTD is defined as highest dose level in which 6 patients have been treated with less than 2 instances of dose limiting toxicity (DLT). DLT assessed during the first course of each cohort (28 days), and refers to a study drug related or possibly related event which meets one of the following criteria using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 4.03.

SECONDARY OUTCOMES:
Response Rate of Carfilzomib When Given With Ibrutinib | Assessed after two 28 day cycles
  Response definitions for measurable disease used from Revised International Workshop Standardized Response Criteria for non-Hodgkin's Lymphoma42. Patients assessed for response after every 2 cycles of therapy. Complete response (CR) defined as complete disappearance of all detectable clinical evidence of disease and disease-related symptoms if present before therapy. Partial response (PR) defined as at least a 50% decrease in sum of the product of the diameters (SPD) of up to six of the largest dominant nodes or nodal masses. Stable disease (SD) determined when participant fails to attain criteria needed for a CR or PR, but does not fulfill those for progressive disease. Progressive disease (PD) considered when lymph nodes measure abnormally, if the long axis is more than 1.5 cm regardless of the short axis. If lymph node has a long axis of 1.1 to 1.5 cm, it should only be considered abnormal if its short axis is more than 1.0.

CONTACTS AND LOCATIONS:
Overall Officials: Hun J. Lee, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org